CLINICAL TRIAL: NCT06515210
Title: Clinical Profiling of Anti-inflammatory Fibre Supplements in Patients With Ulcerative Colitis: Towards Personalized Complementary Strategies.
Brief Title: Personalized Anti-Inflammatory Fibres in Ulcerative Colitis
Acronym: PAIF-UC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Weston Family Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00137948
Record Dates: First submitted 2024-07-10; First posted 2024-07-23 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Ulcerative Colitis
Keywords: inflammatory bowel disease; ulcerative colitis; dietary fibre; gut microbiome
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Gum Arabic; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, parallel-arm, placebo-controlled, six-week clinical trial, with optional 6-week extension for participants in whom the primary outcome is achieved.
Who Masked: Participant, Investigator
Masking Description: The study is double-blinded. The fibre supplements are provided in individual daily sachets, packaged and code-labelled by researchers not involved in data analysis or patient care to ensure double-blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acacia Gum (Experimental): Acacia gum is a dietary fibre with low-viscosity and is fermentable.
  Female participants consume 12.5 grams each day for the first two days of the intervention, then consume 25 grams each day for the rest of the six-week intervention.
  Male participants consume 17.5 grams each day for the first two days of the intervention, then consume 35 grams each day for the rest of the six-week intervention.
  Those participants who voluntarily extend their treatment for an additional six weeks will continue with consuming the full dose daily.
  Interventions: Dietary Supplement: Acacia Gum
- Microcrystalline Cellulose (Experimental): Microcrystalline cellulose is a dietary fibre that is non-viscous and and non-fermentable.
  Female participants consume 12.5 grams each day for the first two days of the intervention, then consume 25 grams each day for the rest of the six-week intervention.
  Male participants consume 17.5 grams each day for the first two days of the intervention, then consume 35 grams each day for the rest of the six-week intervention.
  Those participants who voluntarily extend their treatment for an additional six weeks will continue with consuming the full dose daily.
  Interventions: Dietary Supplement: Microcrystalline Cellulose
- Maltodextrin (Placebo Comparator): Maltodextrin is a digestible carbohydrate. It is provided in isocaloric doses to the dietary fibres.
  Female participants consume 6.3 grams each day for the first two days of the intervention, then consume 12.5 grams each day for the rest of the six-week intervention.
  Male participants consume 8.8 grams each day for the first two days of the intervention, then consume 17.5 grams each day for the rest of the six-week intervention.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Acacia Gum — Participants (n=23) incorporate the fibre supplement into their usual diet daily.
  Other Names: AGRI-SPRAY ACACIA® R, Agrigum International
  Arms: Acacia Gum
Dietary Supplement: Microcrystalline Cellulose — Participants (n=23) incorporate the fibre supplement into their usual diet daily.
  Other Names: MICROCEL® MC-12, ROQUETTE
  Arms: Microcrystalline Cellulose
Dietary Supplement: Placebo — Participants (n=23) incorporate the placebo into their usual diet daily.
  Other Names: GLUCIDEX® IT 19 - MALTODEXTRIN, ROQUETTE
  Arms: Maltodextrin

SUMMARY:
The goal of this clinical trial is to determine the clinical effects of two different dietary fibre supplements, acacia gum (AG) and microcrystalline cellulose (MCC), in patients with ulcerative colitis. The main question it aims to answer is: Can the fibre supplements reduce gut inflammation (fecal calprotectin)?

Researchers will compare AG and MCC to a placebo (a look-alike substance that contains no fibre) to see if the fibre supplements improve inflammation in ulcerative colitis.

Participants will add their assigned fibre supplement or placebo to their usual diet daily for 6 weeks. They will visit the clinic at baseline, week 3, and week 6 to provide samples (stool, blood) and complete various questionnaires.

DETAILED DESCRIPTION:
Prevalence and incidence of inflammatory bowel diseases (IBD), including ulcerative colitis (UC), is rising rapidly in Canada and the rates are amongst the highest globally (Crohn's and Colitis Canada, 2023). UC is a chronic disease characterized by colonic inflammation, often inadequately managed in the long-term with immunosuppressive medications that can increase risk of infections and malignancies (Kayal & Shah, 2019). Alternative, complementary strategies are, therefore, necessary to improve patient outcomes.

A potential target for such strategies may be the gut microbiome, which can predict failure of standard therapy in pediatric UC (Michail et al., 2012). Putative, pro-inflammatory microbes are enriched in patients with IBD compared to healthy controls and disease phenotypes can be transferred via microbiome transplantation into germ-free mice (Nagao-Kitamoto et al., 2016; Birtton et al., 2019), suggesting a causal role of the gut microbiome in IBD. Fibre-based treatments for UC have been proposed and tested for UC but results are mixed, quite modest in many cases, and many gaps remain in defining the most appropriate clinical approach (Di Rosa et al., 2022; Limketkai et al, 2020).

Dietary fibre has great potential as a safe, complementary, microbiome-targeted treatment strategy to reduce inflammation in UC. Food supplementation with fermentable fibres alters microbiome composition (So et al., 2018) and increases microbial production of bioactive metabolites like short-chain fatty acids (SCFAs) that can attenuate inflammation (Parada Venegas et al., 2019; Levine et al., 2018). Provision of growth substrates in the form of fibre also enhances gut barrier function by decreasing mucus degradation, thus reducing bacterial encroachment and immune activation that may drive inflammation (Desai et al., 2016; Earle et al., 2015). However, specific fibre structures elicit distinct health effects due to differences in physicochemical properties (Gill et al., 2020). Therefore, important open questions remain, such as which fibres and physicochemical properties are most beneficial in the context of UC, and are their effects microbiome-dependent?

Hypothesis: Acacia gum (AG; soluble and fermentable fibre) and microcrystalline cellulose (MCC; insoluble and non-fermentable fibre) will decrease gut inflammation in patients with UC, but through different mechanisms given their differences in fermentability.

The overall goal of this study is to determine the clinical effects of AG and MCC in patients with UC, using normalization of FCP as the primary outcome.

Voluntary trial extension: Participants in whom the primary outcome has been achieved at week 6 will be invited to participate in an optional (completely voluntary) extension of the trial and continue their assigned treatment for an additional six weeks. This will allow for exploratory assessment of longer-term efficacy of the fibres (primary and secondary outcomes assessed again at week 12). Apart from the planned study, if a clinical decision is made by the patient and physician to perform sigmoidoscopy or colonoscopy (which is justified in many cases), bio samples and data from these procedures will be collected if patients agree. The procedure will not be a research procedure, but the patients will be approached and consented for bio sample collection. The optional extension will advantageously provide further biological insights into the effects of the fibres and can inform future intervention studies.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of ulcerative colitis.
* Measured fecal calprotectin of >250 µg/g at screening.
* Mild disease: Partial Mayo Scoring Index Assessment for UC between 0-4 (adult patients).
* Mild disease: Pediatric UC Activity Index (PUCAI) between 0-34 (pediatric patients).
* Tanner stage 5 for pediatric patients.
* Weight >50kg.
* No changes to IBD-related medications in three months prior to study onset (stable therapy, including use of 5-aminosalicylic acid, biologics, and immunosuppressive medications; some minor adjustments allowed, such as increasing dose for weight change, or change to a compatible/generic treatment).
* Men and women; the latter must be menstruating and using contraceptives.

Exclusion Criteria:

* Inability to provide informed consent.
* Presence of Crohn disease, IBD unclassified, non-IBD bowel conditions (e.g., celiac), or motility disorder.
* Use of systemic antibiotics for more than a week during two months prior to intervention, or any antibiotic use during the intervention.
* Use of probiotic, prebiotic, or fibre supplements in month prior to intervention known to affect the gut microbiome (if these are present in foods, such as yogurt or fermented foods, this will be allowed).
* Chronic use of laxatives or stool softeners.
* History of abdominal surgery, including appendectomy.
* Pregnancy or intention of the patient to become pregnant during the study period.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in fecal calprotectin | Week 3 and Week 6 (and week 12, if applicable)
  Calprotectin will be analyzed in fecal samples. Clinically-relevant reductions are defined as levels <150 µg/g or reduced by at least 50% from baseline.

SECONDARY OUTCOMES:
Changes in disease activity | Week 3 and Week 6 (and week 12, if applicable)
  Scores obtained from either the Partial Mayo Scoring Index Assessment for adult participants or the Pediatric Ulcerative Colitis Activity Index for pediatric participants.
Changes in fecal microbiome composition | Week 3 and Week 6 (and week 12, if applicable)
  Fecal microbiome composition will be analyzed using whole metagenome sequencing to measure changes at different taxonomic levels (e.g. genus, species).
Changes in function of the fecal microbiome | Week 3 and Week 6 (and week 12, if applicable)
  Fecal microbiome functions will be analyzed using whole metagenome sequencing to measure changes in enzymes and pathways encoded by gut microbiota.
Changes in gut barrier function: fecal zonulin | Week 3 and Week 6 (and week 12, if applicable)
  Fecal samples will be analyzed for changes in zonulin (ng/mg).
Changes in gut barrier function: plasma lipopolysaccharide binding protein | Week 3 and Week 6 (and week 12, if applicable)
  Plasma from blood samples will be analyzed for changes in lipopolysaccharide binding protein (µg/mL).
Changes in fecal short-chain fatty acids | Week 3 and Week 6 (and week 12, if applicable)
  Short-chain fatty acids (acetate, propionate, butyrate, valerate) and branched-chain fatty acids (isovalerate, isobutyrate) will be measured in fecal samples using gas chromatography mass spectrometry (µmol/g).
Changes in fecal bile acids | Week 3 and Week 6 (and week 12, if applicable)
  Bile acid derivatives will be measured in fecal samples using ultrahigh performance liquid chromatography/multiple-reaction monitoring-mass spectrometry (nmol/g).
Changes in fecal pH | Week 3 and Week 6 (and week 12, if applicable)
  Fecal pH will be measured using a pH meter.
Changes in fecal dry mass percentage | Week 3 and Week 6 (and week 12, if applicable)
  Fecal moisture content, or percentage of dry mass, will be measured by drying fecal material overnight in an oven.
Changes in the plasma metabolome | Week 3 and Week 6 (and week 12, if applicable)
  Untargeted metabolomics will be applied to plasma samples via high performance chemical isotope labeling liquid chromatography mass spectrometry platform.
Changes in the plasma inflammatory cytokines | Week 3 and Week 6 (and week 12, if applicable)
  Several inflammatory cytokines (e.g., TNF-α, IL-6) will be analyzed in plasma samples using multiplex, electrochemiluminescence assays.
Changes in routine clinical bloodwork | Week 3 and Week 6 (and week 12, if applicable)
  Routine clinical bloodwork will be performed for patients (e.g., C-reactive protein, liver enzymes, albumin, etc.)
Changes in body weight | Week 3 and Week 6 (and week 12, if applicable)
  Body weight will be measured in kilograms and will be used to calculate body mass index.
Changes in gastrointestinal symptoms | Week 3 and Week 6 (and week 12, if applicable)
  Individual gastrointestinal symptoms will be measured by a gastrointestinal symptom questionnaire (scored on a scale of 0-5; higher scores indicating more symptoms).
Changes in dietary intake | Week 3 and Week 6 (and week 12, if applicable)
  Dietary intake will be measured by 24 hour dietary recalls (using ASA-24).
Changes in patient quality of life | Week 3 and Week 6 (and week 12, if applicable)
  Patient quality of life will be evaluated using the EQ-5D-5L questionnaire.
Need for rescue therapy | Week 3 and Week 6 (and week 12, if applicable)
  Changes to patient therapy regimes (e.g., steroids, dose escalation), inability to complete the study, and adverse events related to the intervention will be monitored and analyzed.

OTHER OUTCOMES:
Biopsies, Brushings, Intestinal Washes, and Endoscopy Scores | Week 12
  In those participants who voluntarily extend their treatment for an additional six weeks, if a clinical decision is made by the patient and physician to perform sigmoidoscopy or colonoscopy, biosamples (biopsies, brushing, and intestinal washes) and data (endoscopy scores) will be collected from these procedures if patients agree. The procedure will not be a research procedure, but the patients will be approached and consented for biosample collection.

CONTACTS AND LOCATIONS:
Overall Officials: Eytan Wine, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared that underlies the results reported after deidentification (text, tables, figures, and appendices). Data will be made available through a safe and secure publicly available data sharing repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication, ending 5 years following publication.
Access Criteria: Anyone who wishes to access the data may do so to achieve aims in the approved proposal and for individual participant data meta-analysis.

REFERENCES:
- [Background] Crohn's and Colitis Canada. Impact of inflammatory bowel disease in Canada. Available from: https://crohnsandcolitisca/About-Us/Resources-Publications/Impact-of-IBD-Report2023.
- [Background] Kayal M, Shah S. Ulcerative Colitis: Current and Emerging Treatment Strategies. J Clin Med. 2019 Dec 30;9(1):94. doi: 10.3390/jcm9010094. PMID 31905945
- [Background] Michail S, Durbin M, Turner D, Griffiths AM, Mack DR, Hyams J, Leleiko N, Kenche H, Stolfi A, Wine E. Alterations in the gut microbiome of children with severe ulcerative colitis. Inflamm Bowel Dis. 2012 Oct;18(10):1799-808. doi: 10.1002/ibd.22860. Epub 2011 Dec 14. PMID 22170749
- [Background] Nagao-Kitamoto H, Shreiner AB, Gillilland MG 3rd, Kitamoto S, Ishii C, Hirayama A, Kuffa P, El-Zaatari M, Grasberger H, Seekatz AM, Higgins PD, Young VB, Fukuda S, Kao JY, Kamada N. Functional Characterization of Inflammatory Bowel Disease-Associated Gut Dysbiosis in Gnotobiotic Mice. Cell Mol Gastroenterol Hepatol. 2016 Mar 3;2(4):468-481. doi: 10.1016/j.jcmgh.2016.02.003. eCollection 2016 Jul. PMID 27795980
- [Background] Britton GJ, Contijoch EJ, Mogno I, Vennaro OH, Llewellyn SR, Ng R, Li Z, Mortha A, Merad M, Das A, Gevers D, McGovern DPB, Singh N, Braun J, Jacobs JP, Clemente JC, Grinspan A, Sands BE, Colombel JF, Dubinsky MC, Faith JJ. Microbiotas from Humans with Inflammatory Bowel Disease Alter the Balance of Gut Th17 and RORgammat+ Regulatory T Cells and Exacerbate Colitis in Mice. Immunity. 2019 Jan 15;50(1):212-224.e4. doi: 10.1016/j.immuni.2018.12.015. PMID 30650377
- [Background] Di Rosa C, Altomare A, Imperia E, Spiezia C, Khazrai YM, Guarino MPL. The Role of Dietary Fibers in the Management of IBD Symptoms. Nutrients. 2022 Nov 11;14(22):4775. doi: 10.3390/nu14224775. PMID 36432460
- [Background] Limketkai BN, Gordon M, Mutlu EA, De Silva PS, Lewis JD. Diet Therapy for Inflammatory Bowel Diseases: A Call to the Dining Table. Inflamm Bowel Dis. 2020 Mar 4;26(4):510-514. doi: 10.1093/ibd/izz297. PMID 31819987
- [Background] So D, Whelan K, Rossi M, Morrison M, Holtmann G, Kelly JT, Shanahan ER, Staudacher HM, Campbell KL. Dietary fiber intervention on gut microbiota composition in healthy adults: a systematic review and meta-analysis. Am J Clin Nutr. 2018 Jun 1;107(6):965-983. doi: 10.1093/ajcn/nqy041. PMID 29757343
- [Background] Parada Venegas D, De la Fuente MK, Landskron G, Gonzalez MJ, Quera R, Dijkstra G, Harmsen HJM, Faber KN, Hermoso MA. Short Chain Fatty Acids (SCFAs)-Mediated Gut Epithelial and Immune Regulation and Its Relevance for Inflammatory Bowel Diseases. Front Immunol. 2019 Mar 11;10:277. doi: 10.3389/fimmu.2019.00277. eCollection 2019. PMID 30915065
- [Background] Levine A, Sigall Boneh R, Wine E. Evolving role of diet in the pathogenesis and treatment of inflammatory bowel diseases. Gut. 2018 Sep;67(9):1726-1738. doi: 10.1136/gutjnl-2017-315866. Epub 2018 May 18. PMID 29777041
- [Background] Desai MS, Seekatz AM, Koropatkin NM, Kamada N, Hickey CA, Wolter M, Pudlo NA, Kitamoto S, Terrapon N, Muller A, Young VB, Henrissat B, Wilmes P, Stappenbeck TS, Nunez G, Martens EC. A Dietary Fiber-Deprived Gut Microbiota Degrades the Colonic Mucus Barrier and Enhances Pathogen Susceptibility. Cell. 2016 Nov 17;167(5):1339-1353.e21. doi: 10.1016/j.cell.2016.10.043. PMID 27863247
- [Background] Earle KA, Billings G, Sigal M, Lichtman JS, Hansson GC, Elias JE, Amieva MR, Huang KC, Sonnenburg JL. Quantitative Imaging of Gut Microbiota Spatial Organization. Cell Host Microbe. 2015 Oct 14;18(4):478-88. doi: 10.1016/j.chom.2015.09.002. Epub 2015 Oct 1. PMID 26439864
- [Background] Gill SK, Rossi M, Bajka B, Whelan K. Dietary fibre in gastrointestinal health and disease. Nat Rev Gastroenterol Hepatol. 2021 Feb;18(2):101-116. doi: 10.1038/s41575-020-00375-4. Epub 2020 Nov 18. PMID 33208922